CLINICAL TRIAL: NCT06884592
Title: Determination of the Incidence of Difficult Intubation and Predictive Factors in Patients Undergoing Nasal Septum Deviation Surgery.
Brief Title: Determination of the Frequency and Predictors of Difficult Intubation in Septoplasty Operations
Status: Recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine OZCAN, Specialist Physician, Başakşehir Çam & Sakura City Hospital
Other Study IDs: NSD2025
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Nasal Septum, Irregular; Nasal Septal Defect; Difficult Airway; Difficult Endotracheal Intubation; Predicted Difficult Airway
Keywords: Septoplasty; Nasal Septum Deviation; Difficult Airway; Predicted Difficult Airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Difficult Airway in Septoplasty: The American Society of Anesthesiologists (ASA) I and II patients (aged 18-65 years) with a medical indication for septoplasty under general anaesthesia (requiring tracheal intubation) due to nasal obstruction caused by a deviated nasal septum.
  Interventions: Procedure: Difficult Intubation

INTERVENTIONS:
Procedure: Difficult Intubation — Determination of difficult intubation, according to the Cormack-Lehane scale, intubation will be considered easy for grade I or II and difficult for grade III or IV. If intubation could not be performed with the Macintosh laryngoscope in three attempts, the next step would be to perform intubation with the videolaryngoscope and the third step would be to place the laryngeal mask airway (LMA). The correct position of the tube in the trachea will be confirmed after intubation, preferably by visual confirmation of the tube passing through the glottic opening, auscultation of the chest with a stethoscope and a normal capnograph. If the LMA attempt fails, the patient will be allowed to awaken, with the final step being ventilation using a face mask and consideration of reversing the muscle relaxant effect with sugammadex (4-5 mg/kg). If intubation fails on the first attempt, an intubation stylet will be used if necessary. The intubation method used, total number of attempts for successful i
  Other Names: Predicted Difficult Airway

SUMMARY:
Deviated septum is among the most prevalent etiologies of nasal obstruction. Congenital or acquired deformities of the nasal septum have been demonstrated to result in partial obstruction of the airflow, thereby causing respiratory distress. Furthermore, studies have indicated a potential correlation between nasal congestion and Obstructive Sleep Apnoea Syndrome (OSAS). It is a well-documented phenomenon that patients suffering from nasal obstruction often exhibit an open mouth during sleep, a condition that has been shown to result in the narrowing of the pharyngeal lumen and the subsequent development of sleep-related breathing disorders, including snoring and sleep apnoea. Surgical intervention to correct a deviated nasal septum (commonly referred to as septoplasty) has been shown to reduce upper airway resistance by enhancing airflow, leading to a reduction in the severity of both snoring and OSAS. Numerous studies have demonstrated a robust correlation between a deviated nasal septum and asymmetric facial growth, including maxillary and mandibular abnormalities. While septoplasty is considered a minor surgical procedure with a low anaesthetic risk, concomitant obstructive sleep apnoea syndrome (OSAS) and facial asymmetry have been demonstrated to be associated with an increased risk of difficult intubation. Consequently, the development of preoperative assessment tests to predict difficult intubation is imperative for effective planning of the necessary preoperative preparation when such complications are anticipated. The present study therefore sought to evaluate the incidence of difficult airway in patients undergoing septoplasty. The secondary aim was to determine the predictive factors associated with difficult airway in patients undergoing septoplasty.

DETAILED DESCRIPTION:
Although septoplasty is a minor surgery with low anaesthetic risk, it is a surgical group in which unpredictable difficult airway is frequently encountered due to anatomical facial deformities in patients. To the best of our knowledge, there are no studies on the incidence of difficult airway and predictive factors associated with difficult airway in septoplasty operations. The objectives of this study are threefold: firstly, to determine the incidence of difficult airway in patients undergoing septoplasty surgery; secondly, to ascertain the predictive factors associated with difficult airway in preoperative evaluation; and thirdly, to reduce the complications that may arise from difficult intubation and ensure patient safety by making the necessary difficult airway preparations in the preoperative period in a timely manner. It is anticipated that the study will not engender any additional risks, as no supplementary interventions or medications will be administered to patients beyond those customary to them.

The prospective cohort (observational) study will include American Society of Anesthesiologists (ASA) I and II patients (aged 18-65 years) with an indication for septoplasty under general anaesthesia (requiring tracheal intubation) due to nasal obstruction caused by nasal septum deviation. Patients with a history of difficult intubation and facial trauma or congenital craniofacial deformity, and patients with difficult mask ventilation during the procedure, will be excluded from this study. Preoperative airway assessment will be performed in all patients using the LEMON protocol for difficult airway prediction. The STOP-BANG questionnaire will be administered to all patients in order to determine the risk of OSAS. The upper lip bite test, a component of the preoperative difficult airway assessment, will be employed.Standard monitoring, encompassing electrocardiography (ECG), noninvasive blood pressure, and peripheral oxygen saturation (SpO2), will be conducted. The induction of anaesthesia will be standardised, comprising midazolam at 0.05 mg kg-1, propofol at 2-3 mg kg-1, fentanyl at 1.5 µg kg-1, and rocuronium at 0.6-1 mg kg-1. Mechanical ventilation will be facilitated using a face mask with 100% oxygen. The use of an oropharyngeal airway will be considered if deemed necessary. Neuromuscular function monitoring is a technique that involves electrical stimulation of a motor nerve and monitoring the response of the muscle innervated by this nerve. This monitoring technique may be employed subsequent to neuromuscular blockade. Importantly, it is used to confirm the adequacy of relaxation after administration of neuromuscular blocking agents.The ratio is monitored, and intubation will be performed at TOF: 0/4. For male patients, Macintosh blades number 3 will be used, and for female patients, Macintosh blades number 4 will be used. All intubation procedures will be performed by an anaesthesiologist specialised in the ENT department. Cormack-Lehane laryngeal appearance grades will be noted during laryngoscopy. The Cormack-Lehane scale will be used to determine the difficulty of intubation as follows: grade I or II will be considered easy, and grade III or IV will be considered difficult. If intubation could not be performed with the Macintosh laryngoscope in three attempts, the subsequent steps would be to perform intubation with the videolaryngoscope and then to place the Laryngeal Mask Airway (LMA). The correct position of the tube in the trachea will be confirmed post-intubation, preferably by visual confirmation of the tube passing through the glottic opening, auscultation of the chest with a stethoscope and a normal capnograph. In the event of failure of the LMA attempt, the patient will be permitted to awaken, with the final step being ventilation using a face mask and consideration of reversing the muscle relaxant effect with sugammadex (4-5 mg/kg). In the event of intubation failure on the first attempt, the use of an intubation stylet will be considered if deemed necessary. The intubation method employed, the total number of attempts for successful intubation, stylet use, optimal external laryngeal manipulation application (cricoid pressure) and oropharyngeal airway placement during face mask ventilation will be recorded. The analysis of these values will contribute to the identification of the incidence of difficult airway in patients with deviated nasal septum and the identification of the most common predictive parameter.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients,
* ASA-I-II
* Between the ages of 18 and 65,
* Difficult intubation and no history of facial trauma or congenital craniofacial deformity
* Patients with easy mask ventilation during the procedure
* Nasal obstruction due to deviated nasal septum,
* Patients who will receive general anaesthesia and undergo septoplasty surgery

Exclusion Criteria:

* Patients without consent
* Not in the appropriate age range,
* Patients who do not receive general anaesthesia and will not undergo septoplasty surgery,
* ASA-IV-V with ,
* Difficult intubation and a history of facial trauma or congenital craniofacial deformity
* Patients with easy mask ventilation during the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with nasal congestion due to deviated nasal septum who will undergo septoplasty surgery under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Cormack-Lehane laryngeal view scale | 3 interventions during procedure
  The anaesthesiologist's assessment is based on the laryngoscopic view of Cormack-Lehane. The Cormack- Lehane test categorises the following grades:
  Grade I: Entire glottis is visible; Grade II: Glottis partially visible; Grade III: Only the epiglottis is visible; Grade IV: Epiglottis also not visible Grade III and IV are considered difficult intubation.

CONTACTS AND LOCATIONS:
Overall Officials: EMINE OZCAN, Anesthesiologist, Principal Investigator — Başakşehir Çam ve Sakura Şehir Hastanesi; HILAL AKÇA, Anesthesiologist, Study Chair — Başakşehir Çam ve Sakura Şehir Hastanesi
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Başakşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying the results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months after publication of the results

REFERENCES:
- [Background] Demet Altun, Achmet Ali, Levent Aydemir, Nil Kırşan, Mukadder Orhan Sungur, Emre Çamcı Determination of the Difficult Intubation Incidence and its Affecting Factors in Patients Undergoing Septal Deviation Surgery Prospective Controlled Trial DOI:10.14744/scie.2019.55477 South.Clin.Ist. Euras.2020;31(1):1-7
- [Background] Dr.Neha Sharma, Dr.Suman Shekhar Tiwari, Dr.Anurag Srivastava, Dr.Prakriti Gupta The preoperative evaluation of risk variables associated with difficult intubation International Journal of Life Sciences Biotechnology and Pharma Research Vol. 12, No. 2, April- June 2023 ISSN: 2250-3137
- [Background] Karakus O, Kaya C, Ustun FE, Koksal E, Ustun YB. [Predictive value of preoperative tests in estimating difficult intubation in patients who underwent direct laryngoscopy in ear, nose, and throat surgery]. Rev Bras Anestesiol. 2015 Mar-Apr;65(2):85-91. doi: 10.1016/j.bjan.2014.05.011. Epub 2014 Nov 28. Portuguese. PMID 25435415
- [Background] Mathangi K, Mathews J, Mathangi CD. Assessment of perioperative difficult airway among undiagnosed obstructive sleep apnoea patients undergoing elective surgery: A prospective cohort study. Indian J Anaesth. 2018 Jul;62(7):538-544. doi: 10.4103/ija.IJA_158_18. PMID 30078857
- See also: The National Center for Biotechnology Information advances science and health by providing access to biomedical and genomic information. And Southern Clinics of Istanbul Eurasia — https://scie.online/jvi.aspx?un=SCIE-55477